CLINICAL TRIAL: NCT02130141
Title: The Effects of Dark Chocolate on Blood Pressure in Mildly Hypertensive Individuals
Brief Title: The Effects of Dark Chocolate on Blood Pressure in Individuals With Mildly Elevated Blood Pressure
Acronym: CHOKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Fazer Group (Industry)
Responsible Party: Principal Investigator, Mikael Fogelholm, Professor, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HY-RAV-FAZ-01
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Blood Pressure
Keywords: cocoa; dark chocolate; hypertension; blood pressure monitoring, ambulatory; flavanols
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dark chocolate, dietary counselling (Experimental): Mildly hypertensive subject will replace their usual snacks with with 50 g dark chocolate daily for a period of 8 weeks.
  Interventions: Dietary Supplement: Dark chocolate
- Dietary counselling (Active Comparator): Usual snacks are limited.
  Interventions: Dietary Supplement: Dark chocolate; Other: Dietary counselling

INTERVENTIONS:
Dietary Supplement: Dark chocolate — Mildly hypertensive subject will replace their usual snacks with with 50 g dark chocolate daily for a period of 8 weeks.
Other: Dietary counselling — Usual snacks are limited.
  Arms: Dietary counselling

SUMMARY:
The evidence linking chocolate with lowered blood pressure has been observed. However, the interventions have been short, at most 4 weeks. The aim of this study is to find out if the habitual consumption of dark chocolate for 8 weeks has an effect on blood pressure. Also, more insight to the mechanisms linking chocolate to individual healt-responses is needed.

ELIGIBILITY:
Inclusion Criteria:

* age 25-65 years
* resting systolic pressure 140-159 mmHg or diastolic blood pressure 90-99 mmHg
* BMI 25.0- 29.9

Exclusion Criteria:

* smoking
* regular medication for hypertension, cardiovascular disease, diabetes or asthma

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in systolic and diastolic blood pressure | 8 weeks
  Usual daily snack is replaced by 50 g dark chocolate for a period of 8 weeks. During the control period, the same usual snack is limited in the diet, but without the replacement with the dark chocolate.

SECONDARY OUTCOMES:
Ambulatory blood pressure | 8 weeks
Blood lipids, inflammation markers, plasma levels of cocoa polyphenols | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Fogelholm, Dr., Principal Investigator — University of Helsinki
Locations (2):
- Finland (2):
  - University of Helsinki, Helsinki, Helsingin Yliopisto
  - Institute of Clinical Medicine, Helsinki, Uusimaa

REFERENCES:
- [Derived] Koli R, Kohler K, Tonteri E, Peltonen J, Tikkanen H, Fogelholm M. Dark chocolate and reduced snack consumption in mildly hypertensive adults: an intervention study. Nutr J. 2015 Aug 22;14:84. doi: 10.1186/s12937-015-0075-3. PMID 26296850